CLINICAL TRIAL: NCT06115135
Title: A Phase 2 Study of Venetoclax in Combination With Isatuximab and Dexamethasone for Relapsed/Refractory Multiple Myeloma Patients With t(11;14)
Brief Title: A Study of Venetoclax in Combination With Isatuximab and Dexamethasone for Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-VID-2022
Record Dates: First submitted 2023-08-11; First posted 2023-11-02 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; MM; RRMM; Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- open-label (Experimental): This is a Phase 2, multicenter, open-label study evaluating the safety and efficacy of venetoclax in combination with isatuximab and dexamethasone among RRMM patients who show the t(11;14) marker and currently show PD and have received at least 3 prior lines of therapy for multiple myeloma. All subjects in Dose Level 0 will receive 1) venetoclax, PO, at 400 mg every day (QD) on Days 1-28 of a 28-day cycle, 2) dexamethasone 40 mg IV, once weekly on Days 1, 8, 15, and 22 of a 28-day cycle where day 8 and 22 doses may be administered PO; and 3) isatuximab 10mg/kg, IV, on Days 1, 8, 15, and 22 of the first 28-day cycle, and then Days 1 and 15 during subsequent 28-day cycles.
  The primary safety analysis will focus on determining the DLTs for the study regimen, and occurrence of AEs throughout the study.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — All subjects in Dose Level 0 will receive 1) venetoclax, PO, at 400 mg every day (QD) on Days 1-28 of a 28-day cycle, 2) dexamethasone 40 mg IV, once weekly on Days 1, 8, 15, and 22 of a 28-day cycle; and 3) isatuximab 10mg/kg, IV, on Days 1, 8, 15, and 22 of the first 28-day cycle, and then Days 1 and 15 during subsequent 28-day cycles.
  Other Names: VENCLEXTA

SUMMARY:
A phase 2 study of venetoclax in combination with isatuximab and dexamethasone for relapsed/refractory multiple myeloma patients with t(11;14)

DETAILED DESCRIPTION:
Despite recent advances in treating MM that have improved outcomes, patients with this B-cell malignancy inevitably become refractory to therapy, and thus, must rely on additional treatment options for long-term management of their disease.

Venetoclax is an oral BCL-2 inhibitor which has been recently demonstrated to show clinical activity for the treatment of MM. The BCL-2 family of proteins are critical regulators of apoptosis which include both anti-apoptotic (e.g. BCL-2, MCL-1 and BCL-XL) and pro-apoptotic (e.g. BAK and BAX) elements. The upregulation of anti-apoptotic proteins has been reported for most cancers, but high BCL-2 levels have been especially prevalent in human lymphoid malignancies including chronic lymphocytic leukemia, for which venetoclax is currently indicated. BCL-2 is also overexpressed especially in the subset of MM patients with t(11;14) translocations, a cytogenetic abnormality found in approximately 20% of MM patients.

Venetoclax as a single agent has been shown to induce apoptosis not only in human MM cell lines and primary MM tumor cell samples, but also specifically in RRMM patients. Clinical activity with single-agent venetoclax was mostly limited to those with (11;14) translocations, with 12 of 14 responses occurring among patients with that cytogenetic marker in the single-agent clinical trial of this BCL-2 inhibitor for patients with RRMM (#NCT01794520) as reported by Kumar et al.7 Resistance to venetoclax as a single agent has been shown to be mediated by MCL-1, with low BCL-2/MCL-1 ratios indicating resistance and high ratios indicating an increased sensitivity to this BCL-2 inhibitor. Furthermore, MCL-1 silencing was shown to heighten sensitivity to BCL-2 inhibitors, and MM xenograft models co-expressing BCL-2 with MCL-1 were resistant to venetoclax.

The therapeutic landscape of MM has evolved even more with the discovery and validation of monoclonal antibodies in the treatment of MM. The first two monoclonal antibody-based therapies to show promising activity for treating MM patients were elotuzumab, which targets SLAMF7, and daratumumab, which targets CD38. A recent phase 1 study showed high response rates among RRMM patients with t(11;14) who were treated with daratumumab, dexamethasone and venetoclax.2 The most recent addition to the collection of the antibody-based therapies is a humanized IgG1 monoclonal antibody that binds selectively to a unique epitope on the human CD38 receptor, isatuximab (SAR-650984). A dose finding phase 2 trial of isatuximab as a single agent was well tolerated and showed clinical activity for heavily pre-treated patients with RRMM.3 Furthermore, a phase 1b study examining combination therapy consisting of isatuximab with lenalidomide and dexamethasone showed promising activity and good tolerability for heavily previously treated patients with RRMM. Based on the results of two phase 3 studies, the antibody has been FDA-approved in combination with pomalidomide or carfilzomib for treating RRMM patients.

Notably, the investigators reported two cases of patients with RRMM who achieved rapid complete remissions to therapy with venetoclax at low doses (100 mg) in combination with bortezomib, dexamethasone and the anti-CD38 antibody daratumumab after failing multiple treatment regimens including bortezomib, dexamethasone and daratumumab. The investigators have recently reported on a larger retrospective study of RRMM patients receiving this combination. The response rate was 80% among those harboring the t(11;14) marker whereas it was only 31% among those lacking this chromosomal translocation. Responses were observed among patients who failed prior anti-CD38 antibody treatments. These results suggest that low doses of venetoclax may help overcome resistance to other anti-MM agents for the treatment of RRMM patients especially those with the t(11;14) chromosomal marker. Therefore, in this phase 2 trial, The investigators will evaluate the safety and efficacy of isatuximab, venetoclax and dexamethasone for treating patients with RRMM and show the t(11;14) marker.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be eligible to enroll in this study.

1.Has a diagnosis of MM based on standard criteria as follows: Myeloma Criteria: Must be At least 1 of 2

1. Clonal bone marrow plasma cells >10%
2. Biopsy-proven bony or extramedullary plasmacytoma

Active Myeloma criteria: Must Meet At Least ONE of the Following:

Meet at least one of the sub-criteria for #1 Evidence of End Organ Damage (a, b, c, or d), OR Meet sub-criteria #2. 60% or greater bone marrow plasma cells, OR Meet sub-criteria #3 Serum free light chain ratio, OR Meet sub-criteria #4 More than one focal lesion on MRI > 5mm in size.

1. Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically

   1. Hypercalcemia: serum calcium >0.25 mmol/L (>1mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11mg/dL)
   2. Renal insufficiency: creatinine clearance <40 mL per minute or serum creatinine >177mol/L (>2mg/dL)
   3. Anemia: hemoglobin value of >20g/L below the lowest limit of normal, or a hemoglobin value <100g/L
   4. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET/CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement
2. 60% or greater clonal plasma cells on bone marrow examination
3. Serum involved / uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved light chain is at least 100 mg/L (a patient's involved free light chain either kappa or lambda is the one that is above the normal reference range; the uninvolved free light chain is the one that is typically in, or below, the normal range)
4. More than one focal lesion on MRI that is at least 5mm or greater in size The patient must have met the criteria for Active Myeloma at some stage following the diagnosis of Myeloma. Source documentation for both Myeloma and Active Myeloma will be required.

2. Currently has MM with measurable disease, defined as:

1. a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or urine monoclonal protein levels of at least 200 mg/24 hours
2. for patients without measurable serum and urine M-protein levels, an involved SFLC > 100 mg/L or abnormal SFLC ratio
3. for patients with IgD MM, a monoclonal immunoglobulin IgD of at least 1500 mg/L or meet other measurable disease eligibility criteria

   3. Show the (11;14), as demonstrated by FISH or cytogenetic analysis at screening or at any point prior to screening. If performed more than 45 days prior, it should be repeated at the investigator's discretion.

   4. Absolute neutrophil count ≥ 1.5 x 109/L 5. Platelet count ≥ 75 x 109/L 6. Hemoglobin ≥ 8.0 g/dL within 21 days prior to enrollment. 7. Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/minute as calculated by Cockcroft-Gault method 8. Total bilirubin levels ≤ 2.0 mg/dL (normal levels) 9. AST (SGOT) and ALT (SGPT) ≤ 2 x ULN 10. Serum potassium 3.0-5.5 mEq/L 11. Female of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting and must either commit to continued abstinence from heterosexual intercourse or use acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, and at least 28 days before she starts taking treatment drugs. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Contraception measures should be continued for 3 months following the treatment completion.

   †A FCBP (female of childbearing potential) is a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months 12. Eastern Cooperative Oncology Group (ECOG) performance score less than or equal to 2 13. Participant must have received at least 1 prior line of therapy for multiple myeloma, including a proteasome inhibitor, lenalidomide, and glucocorticosteroids but not necessarily in one treatment regimen 14. Participant currently has documented progressive MM per IMWG criteria

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Participant has a history of intolerability to any of the study drugs
2. Participant has any of the following conditions: amyloidosis, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), known human immunodeficiency viral (HIV) infection, active hepatitis B or C infection based on blood screen tests, significant cardiovascular disease, including uncontrolled angina, severe or uncontrolled arrhythmia, recent myocardial infarction within 6 months of screening, or congestive heart failure New York Heart Association (NYHA) Class greater than or equal to 3, Major surgery within 4 weeks prior to screening, acute infections requiring parenteral therapy (antibiotic, antifungal, or antiviral) within 14 days prior to screening, uncontrolled diabetes or uncontrolled hypertension within 14 days prior to screening, any other medical condition that, in the opinion of the Investigator, would adversely affect the participant's participation in the study
3. Participant has a history of other active malignancies, including myelodysplastic syndrome (MDS), within the past 3 years prior to study entry, with the following exceptions: previous malignancy with no evidence of disease confined and surgically resected (or treated with other modalities) with curative intent and unlikely to impact survival during the duration of the study
4. If participant had prior allogeneic stem cell transplant (SCT), participant has evidence of ongoing graft-versus-host disease (GvHD)
5. Participants that are pregnant or breast feeding
6. Participants with hypersensitivity to any study medications and/or their excipients
7. Treatment with an anti-CD38 antibody (daratumumab or isatuximab) within the last 3 weeks
8. For those patients treated with an anti-CD38 antibody (daratumumab or isatuximab), alone or in combination, without achieving a best response of at least MR
9. Treatment with venetoclax
10. Treatment with any of the following prior to the first dose of study drug:

    1. Chemotherapy within 3 weeks of starting study drugs
    2. Corticosteroids (>20 mg per day prednisone or equivalent) within 3 weeks of starting study drugs
    3. Immunotherapy, antibody therapy, immunomodulatory agents, or proteasome inhibitors within 3 weeks of starting study drugs
    4. Extensive radiation therapy within 28 days of starting study drugs. Receipt of localized radiation therapy does not preclude enrollment
    5. Use of any other experimental drug or therapy within 28 days of starting study drugs
    6. Moderate or strong cytochrome P450 3A (CYP3A) inhibitors or inducers within 7 days of starting study drugs
11. Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

    1. Grapefruit or grapefruit products
    2. Seville oranges (including marmalade containing Seville oranges)
    3. Star fruit
12. Additional prior and concomitant therapy excluded and cautionary medications:

    a. Excluded: i. Anticancer therapies including chemotherapy, radiotherapy, or other investigational therapy, including targeted small molecule agents: Excluded 5 half-lives prior to first dose and throughout venetoclax administration ii. Biologic agents (e.g., monoclonal antibodies) for anti-neoplastic intent: Excluded 21 days prior to first dose and throughout venetoclax administration
13. Cautionary during the study:

    1. Strong and Moderate CYP3A inhibitors: Exclude during ramp-up phase and consider alternative medications. If the subject requires use of these medications at the cohort designated dose, use with caution and reduce the venetoclax dose by 50% for moderate inhibitors and at least 75% for strong inhibitors during co-administration. After discontinuation of CYP3A inhibitor, wait for 2 to 3 days before venetoclax dose is increased back to the initial maintenance/target dose.
    2. Strong and Moderate CYP3A inducers: Exclude during ramp-up phase and consider alternative medications. If the subject requires use of these medications at the cohort designated dose, use with caution and contact medical monitor for guidance.
    3. Additional: Warfarin, P-gp substrates, BCRP substrates, OATP1B1/1B3 substrates, P-gp inhibitors, BCRP inhibitors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | [Time Frame: 54 months]
  Safety will be measured by counting the occurrence of adverse events throughout the study, graded via Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 criteria
Overall response rate (ORR) as a measure of efficacy | [Time Frame: 54 months]
  To assess the overall response rate (ORR = CR + VGPR + PR)
Clinical benefit rate (CBR) as a measure of efficacy | [Time Frame: 54 months]
  (CBR = CR + VGPR + PR + MR)

SECONDARY OUTCOMES:
Assessment of the time to progression as a measure of efficacy (TTP) | [Time Frame: 54 months]
  Time to progression, defined as the time (in months) from the initiation of therapy to progressive disease.Time to progression, defined as the time (in months) from the initiation of therapy to progressive disease.
Progression Free Survival (PFS) | [Time Frame: 54 months]
  Progression-free survival will be measured in months as the time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
Time to first response (TTFR) | [Time Frame: 54 months]
  Time to first response (TTFR), defined as the time from the initiation of therapy to the first evidence of confirmed clinical benefit defined as > MR including patients who achieved a CR, VGPR, PR, or MR
Duration of response (DOR) | [Time Frame: 54 months]
  Duration of response, defined as the time (in months) from the first response to progressive disease
Overall survival (OS) | [Time Frame: 54 months]
  Overall survival, defined as the time (in months) from initiation of therapy to death from any cause or last follow-up visit

OTHER OUTCOMES:
Biomarker (sBCMA) screening for all patients | [Time Frame: 54 months]
  In this study, we will assess the serum levels of a new serum biomarker for MM, BCMA. It is a tumor necrosis factor receptor family member that is expressed on the surface of normal and malignant B-cells, including MM cells. Serum (s)BCMA levels have been shown to be elevated among MM patients with progressive disease and low among those responding to treatment. In addition to correlating with clinical status, baseline sBCMA levels have been shown to predict PFS and OS. Changes in its levels also mirror those that occur in M protein levels.

CONTACTS AND LOCATIONS:
Overall Officials: James Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (2):
- United States (2):
  - Berenson Cancer Center, West Hollywood, California
  - Nebraska Cancer Specialists, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Bahlis NJ, Baz R, Harrison SJ, Quach H, Ho SJ, Vangsted AJ, Plesner T, Moreau P, Gibbs SD, Coppola S, Yang X, Al Masud A, Ross JA, Bueno O, Kaufman JL. Phase I Study of Venetoclax Plus Daratumumab and Dexamethasone, With or Without Bortezomib, in Patients With Relapsed or Refractory Multiple Myeloma With and Without t(11;14). J Clin Oncol. 2021 Nov 10;39(32):3602-3612. doi: 10.1200/JCO.21.00443. Epub 2021 Aug 13. PMID 34388020
- [Background] Touzeau C, Le Gouill S, Mahe B, Boudreault JS, Gastinne T, Blin N, Caillon H, Dousset C, Amiot M, Moreau P. Deep and sustained response after venetoclax therapy in a patient with very advanced refractory myeloma with translocation t(11;14). Haematologica. 2017 Mar;102(3):e112-e114. doi: 10.3324/haematol.2016.160408. Epub 2017 Jan 5. No abstract available. PMID 28057737
- [Background] Martin T, Baz R, Benson DM, Lendvai N, Wolf J, Munster P, Lesokhin AM, Wack C, Charpentier E, Campana F, Vij R. A phase 1b study of isatuximab plus lenalidomide and dexamethasone for relapsed/refractory multiple myeloma. Blood. 2017 Jun 22;129(25):3294-3303. doi: 10.1182/blood-2016-09-740787. Epub 2017 May 8. PMID 28483761
- [Background] Attal M, Richardson PG, Rajkumar SV, San-Miguel J, Beksac M, Spicka I, Leleu X, Schjesvold F, Moreau P, Dimopoulos MA, Huang JS, Minarik J, Cavo M, Prince HM, Mace S, Corzo KP, Campana F, Le-Guennec S, Dubin F, Anderson KC; ICARIA-MM study group. Isatuximab plus pomalidomide and low-dose dexamethasone versus pomalidomide and low-dose dexamethasone in patients with relapsed and refractory multiple myeloma (ICARIA-MM): a randomised, multicentre, open-label, phase 3 study. Lancet. 2019 Dec 7;394(10214):2096-2107. doi: 10.1016/S0140-6736(19)32556-5. Epub 2019 Nov 14. PMID 31735560
- [Background] Moreau P, Dimopoulos MA, Mikhael J, Yong K, Capra M, Facon T, Hajek R, Spicka I, Baker R, Kim K, Martinez G, Min CK, Pour L, Leleu X, Oriol A, Koh Y, Suzuki K, Risse ML, Asset G, Mace S, Martin T; IKEMA study group. Isatuximab, carfilzomib, and dexamethasone in relapsed multiple myeloma (IKEMA): a multicentre, open-label, randomised phase 3 trial. Lancet. 2021 Jun 19;397(10292):2361-2371. doi: 10.1016/S0140-6736(21)00592-4. Epub 2021 Jun 4. PMID 34097854
- [Background] Rahbari KJ, Nosrati JD, Spektor TM, Berenson JR. Venetoclax in Combination With Bortezomib, Dexamethasone, and Daratumumab for Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2018 Sep;18(9):e339-e343. doi: 10.1016/j.clml.2018.06.003. Epub 2018 Jun 18. No abstract available. PMID 30033209
- [Background] Regidor B, Goldwater MS, Wang J, Bujarski S, Swift R, Eades B, Emamy-Sadr M, Eshagian S, Schwartz G, Spektor TM, Berenson JR. Low dose venetoclax in combination with bortezomib, daratumumab, and dexamethasone for the treatment of relapsed/refractory multiple myeloma patients-a single-center retrospective study. Ann Hematol. 2021 Aug;100(8):2061-2070. doi: 10.1007/s00277-021-04555-3. Epub 2021 May 14. PMID 33987683
- [Background] Smith ML, Newland AC. Treatment of myeloma. QJM. 1999 Jan;92(1):11-4. doi: 10.1093/qjmed/92.1.11. PMID 10209667